CLINICAL TRIAL: NCT03389945
Title: Dural Puncture Epidural For Early Labor Analgesia: A Randomized Comparison Between 27- and 25-Gauge Pencil Point Spinal Needles.
Brief Title: Different Spinal Needles Sizes and Dural Puncture Epidural For Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Felipe Contreras Godoy, Clinical Instructor, Department of Anesthesia, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 922/17
Record Dates: First submitted 2017-12-14; First posted 2018-01-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Labor Pain; Epidural Analgesia
Keywords: Labor analgesia; Dural puncture epidural; Postdural puncture headache; Neuraxial analgesia
MeSH Terms: conditions — Labor Pain; Post-Dural Puncture Headache

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25G Dural Puncture Epidural Block (Active Comparator): Patients will receive a dural puncture epidural block with a 25 gauge spinal needle.
  Interventions: Procedure: 25G Dural Puncture Epidural Block
- 27G Dural Puncture Epidural Block (Experimental): Patients will receive a dural puncture epidural block with a 27 gauge spinal needle.
  Interventions: Procedure: 27G Dural Puncture Epidural Block

INTERVENTIONS:
Procedure: 25G Dural Puncture Epidural Block — Dural puncture epidural analgesia using a 25G pencil point spinal needle at a lumbar interspace.
  Then 20ml of bupivacaine 0.125% + fentanyl 2ug/ml will be injected in the epidural space.
  Arms: 25G Dural Puncture Epidural Block
Procedure: 27G Dural Puncture Epidural Block — Dural puncture epidural analgesia using a 27G pencil point spinal needle at a lumbar interspace.
  Then 20ml of bupivacaine 0.125% + fentanyl 2ug/ml will be injected in the epidural space.
  Arms: 27G Dural Puncture Epidural Block

SUMMARY:
The rationale behind the dural puncture epidural (DPE) technique lies in the fact that a dural perforation with a spinal needle purportedly creates a conduit for accelerated translocation of local anesthetics from the epidural to the subarachnoid space. When compared with conventional epidural block, it provides improved sacral block and onset of analgesia.

Despite the benefits associated, the supportive literature remains scarce. No trial has determined if similar results could be obtained with a smaller needle.

In this trial, DPE using 25- and 27-gauge (G) spinal needles are compared. The main outcome will be the time required to obtain a pain score ≤ 1 using a 0-10 numeric rating scale (NRS). The hypothesis is that that both needle sizes will result in similar onset times and therefore designing the current study as an equivalence trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant woman
* singleton and vertex presentation
* 37-42 weeks of gestational age
* active labor with cervical dilation < 5cm
* body mass index between 20 and 35 kg/m2
* desired labor epidural analgesia

Exclusion Criteria:

* adults who are unable to give their own consent
* presence of any pregnancy-related disease (e.g., gestational hypertension, preeclampsia, gestational diabetes)
* known fetal anomalies
* increased risk of cesarean delivery (e.g., previous uterine rupture, previous cesarean delivery)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or partial prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to LA
* prior sacral or lumbar spine surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-13 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Time to pain ≤ 1 on NRS (0-10) | Up to 30 minutes after local anesthetic injection
  Time elapsed between the end of local anesthetic injection and achievement of pain ≤ 1 on the NRS (measured every 2 minutes)

SECONDARY OUTCOMES:
Gestational age | 42 weeks
  Gestational age at the time of recruitment
Obstetric history | At the time of recruitment
  Number of previous pregnancies and deliveries
Type of labor | At the time of delivery
  Spontaneous versus induced labor
Oxytocin dose | At the time of DPE
  Oxytocin infusion/dose at time of DPE
Cervical dilation | At the time of DPE
  Cervical dilation at the time of DPE
State of membrane | At the time of DPE
  Intact versus ruptured membrane at the time of DPE
Pre-DPE level of pain | Immediate before DPE
  Evaluated with a NRS from 0 to 10
Amount of IV fluids | 24 hours
  Total intravenous fluid received during labor (from admission to the obstetric suite up to delivery)
Intervertebral level of puncture | At the time of DPE
  Lumbar interspace where DPE was successfully performed
Number of DPE attempts | 1 hour
  Number of attempts for successful DPE
Incidence of accidental dural puncture | 1 hour
  Incidence of accidental dural puncture with the epidural Tuohy needle
Performance time | 1 hour
  Temporal interval between skin disinfection and epidural catheter fixation to the skin
Sensory block height | Up to 30 minutes after local anesthetic injection
  Sensory block height at 30 minutes after local anesthetic injection
Bilateral S2 sacral root block | Up to 30 minutes after local anesthetic injection
  Measured every 2 minutes after local anesthetic injection
Presence of motor block | Up to 30 minutes after local anesthetic injection
  Evaluated using a modified Bromage score
Number of epidural top-ups during labor | After DPE up to delivery
  Number of extra doses of local anesthetic given after DPE up to delivery
Type of delivery | Delivery
  Incidence of Cesarean section, normal delivery, and instrumented delivery
Incidence of epidural catheter adjustment or replacement | After DPE up to delivery
  Necessity of adjustment or replacement of the epidural catheter
DPE side effects | After DPE up to delivery
  Incidence of nausea, pruritus, hypotension
Fetal-Uterine assessment | Before and up to 1 hour after DPE
  Frequency of contractions, uterine tonus, fetal heart rate tracing
Tocolysis requirement | Up to 1 hour after DPE
  Necessity to administer a tocolytic agent after DPE
Apgar scores | At 1 and 5 minutes after delivery
  Assessment of newborn condition
DPE complications | After DPE up to 7 days postpartum
  Incidence of post dural puncture headache, back pain, paresthesia and motor deficit
Epidural blood patch incidence | Up to 1 week of followup
  Necessity of performing of a blood patch to relieve post dural puncture headache symptoms

OTHER OUTCOMES:
Demographic data | At the time of recruitment
  Age, height, weight, BMI

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan
  - Hospital La Florida, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suzuki N, Koganemaru M, Onizuka S, Takasaki M. Dural puncture with a 26-gauge spinal needle affects spread of epidural anesthesia. Anesth Analg. 1996 May;82(5):1040-2. doi: 10.1097/00000539-199605000-00028. PMID 8610864
- [Background] Cappiello E, O'Rourke N, Segal S, Tsen LC. A randomized trial of dural puncture epidural technique compared with the standard epidural technique for labor analgesia. Anesth Analg. 2008 Nov;107(5):1646-51. doi: 10.1213/ane.0b013e318184ec14. PMID 18931227
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Background] Tran DQ, Van Zundert TC, Aliste J, Engsusophon P, Finlayson RJ. Primary Failure of Thoracic Epidural Analgesia in Training Centers: The Invisible Elephant? Reg Anesth Pain Med. 2016 May-Jun;41(3):309-13. doi: 10.1097/AAP.0000000000000394. PMID 27035462
- [Background] Thomas JA, Pan PH, Harris LC, Owen MD, D'Angelo R. Dural puncture with a 27-gauge Whitacre needle as part of a combined spinal-epidural technique does not improve labor epidural catheter function. Anesthesiology. 2005 Nov;103(5):1046-51. doi: 10.1097/00000542-200511000-00019. PMID 16249679
- [Background] Landau R, Ciliberto CF, Goodman SR, Kim-Lo SH, Smiley RM. Complications with 25-gauge and 27-gauge Whitacre needles during combined spinal-epidural analgesia in labor. Int J Obstet Anesth. 2001 Jul;10(3):168-71. doi: 10.1054/ijoa.2000.0834. PMID 15321605
- [Background] Beilin Y, Zahn J, Bernstein HH, Zucker-Pinchoff B, Zenzen WJ, Andres LA. Treatment of incomplete analgesia after placement of an epidural catheter and administration of local anesthetic for women in labor. Anesthesiology. 1998 Jun;88(6):1502-6. doi: 10.1097/00000542-199806000-00013. PMID 9637643
- [Derived] Contreras F, Morales J, Bravo D, Layera S, Jara A, Riano C, Pizarro R, De La Fuente N, Aliste J, Finlayson RJ, Tran DQ. Dural puncture epidural analgesia for labor: a randomized comparison between 25-gauge and 27-gauge pencil point spinal needles. Reg Anesth Pain Med. 2019 May 22:rapm-2019-100608. doi: 10.1136/rapm-2019-100608. Online ahead of print. PMID 31118278